CLINICAL TRIAL: NCT06923735
Title: Nutrition Apps in Occupational Healthcare (Pilot Study of the FOODNUTRI Project)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 262/2024
Record Dates: First submitted 2025-03-24; First posted 2025-04-11 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Occupational Diseases; Overweight and Obesity; Dyslipidemias; Hypertension; Diabete Type 2; Cardiovascular Diseases; Diet, Healthy; Diet Habit; Food Selection
MeSH Terms: conditions — Occupational Diseases; Overweight; Obesity; Dyslipidemias; Hypertension; Diabetes Mellitus, Type 2; Cardiovascular Diseases; Feeding Behavior; Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Treatment as usual in the occupational healthcare.
- Intervention (Experimental): Utilization of the nutrition apps in the occupational healthcare.
  Interventions: Other: Utilization of the Finnish Nutrition Navigator and the Finnish Nutrition Path

INTERVENTIONS:
Other: Utilization of the Finnish Nutrition Navigator and the Finnish Nutrition Path — Participant fills in the food intake questionnaire of the Finnish Nutrition Navigator and receives an automated feedback on the diet before the visit to the occupational healthcare. At the visit, the information about the quality of diet can be utilized with the occupational healthcare professional. The client can utilize the self-care path (the Finnish Nutrition Path) for possible dietary changes independently or with the professional.
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate (1) the user experiences and usability of the nutrition apps (the Finnish Nutrition Navigator and the Finnish Nutrition Path) in occupational health care from the perspective of both professionals and customers, (2) the impact on diet, eating behavior, perceived well-being (perceived state of health, quality of life, work and functional ability) and anthropometric indicators compared to treatment as usual, and (3) cost-effectiveness of using the nutrition apps.

DETAILED DESCRIPTION:
For the occupational healthcare customer, the study will include two visits to the occupational healthcare: at baseline and after a 12-week follow-up. First, all volunteer participants enrolled in the study will belong to the control group and they will get the treatment as usual. Their weight, waist circumference, and blood pressure are measured at the visit and they are asked to answer a digital research questionnaire at both baseline and follow-up.

The rest of the volunteer participants enrolled in the study will belong to the intervention group. Before the visit at the occupational healthcare, they are asked to fill in the Finnish Nutrition Navigator and to read the automated feedback about the diet quality. The Finnish Nutrition Path can help in the dietary goal setting and it can be utilized together with the professional or independently. In addition, also weight, waist circumference, and blood pressure are measured at the visit and the participant is asked to answer a digital research questionnaire. The same procedure is done at both baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Employee of the certain employer
* Coming to the medical examination for employees whose work presents a special risk of illnessa OR coming to the dietitian because of dyslipidemia, high blood pressure, weight loss, weight management, type 2 diabetes, cardiovascular disease
* Understands written Finnish

Exclusion Criteria:

* Pregnancy
* Eating disorder
* Severe challenges with diet (e.g., malabsorption, very restrictive diet due to several food allergies or other reasons)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in diet quality | 12 weeks
  Healthy Diet Index (HDI) total score (range 0 - 100) and the seven sub scores: Meal pattern (range 0 - 10), Grains (range 0 - 20), Fruit and vegetables (range 0 - 20), Fats (range 0 - 15), Fish and meat (range 0 - 10), Dairy (range 0 - 10), and Snacks and treats (range 0 - 15). Higher scores mean better diet quality.
User experiences of the apps | Baseline and follow-up (12 weeks)
  Self-created questions.

SECONDARY OUTCOMES:
Change in weight | 12 weeks
  Measured weight in kilograms.
Change in BMI | 12 weeks
  Measured weight and self-reported height will be combined to report BMI in kg/m^2.
Change in waist circumference | 12 weeks
  Measured waist circumference in centimeters.
Change in blood pressure | 12 weeks
  Measured systolic and diastolic blood pressures in mmHg.
Change in eating behavior | 12 weeks
  Questionnaire ecSatter Inventory 2.0TM, ecSI 2.0TM: Total score range 0 - 48 and the four subscales: Eating Attitudes (range 0 - 18), Contextual Skills (range 0 - 15), Food Acceptance (range 0 - 9), and Internal Regulation (range 0 - 6). Higher scores mean better eating competence.
Change in other lifestyle factors | 12 weeks
  Questionnaire: short questions about physical activity, sleep, and smoking.
Measures related to the general effectiveness | 12 weeks
  Questionnaire: questions about perceived health and well-being, quality of life, work productivity and activity impairment, consumer health activation, and life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Marjukka Kolehmainen, Prof., Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No